CLINICAL TRIAL: NCT04392349
Title: Clinical Study - ES 900 - 2020-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haag-Streit AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1023707
Record Dates: First submitted 2020-05-11; First posted 2020-05-18 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cataract; Keratoconus
Keywords: Optical Biometry; Corneal Topography
MeSH Terms: conditions — Cataract; Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NORMAL (Other): Normal group includes eyes with healthy cornea.
  Interventions: Device: Haag-Streit EYESTAR 900; Device: Tomey CASIA 2; Device: Oculus PENTACAM HR; Device: Zeiss ATLAS 9000
- IRREGULAR (Other): Irregular goup includes eyes with irregular astigmatism or corneal scarring.
  Interventions: Device: Haag-Streit EYESTAR 900; Device: Tomey CASIA 2; Device: Oculus PENTACAM HR; Device: Zeiss ATLAS 9000

INTERVENTIONS:
Device: Haag-Streit EYESTAR 900 — The EYESTAR 900 is a new device developed by HAAG-STREIT AG which utilises Optical Coherence Tomography (OCT) for quantitative measurements of the geometry of the eye. As a successor to the LENSTAR 900, it represents the most recent in a series of successful biometry devices.
Device: Tomey CASIA 2 — The CASIA2 is a testing application for Cataract / Glaucoma / Cornea Surgery already established on the market. It is a representative device for measurement of anterior and posterior corneal curvature (anterior and posterior corneal topography) by optical coherence tomography, and for measurement of crystalline lens tilt by optical coherence tomography.
Device: Oculus PENTACAM HR — The Pentacam HR is a high-resolution rotating Scheimpflug camera system for anterior segment analysis already established on the market. It is used as representative device for advanced anterior segment analysis such as anterior and posterior corneal topography and corneal pachymetry.
Device: Zeiss ATLAS 9000 — ATLAS is a corneal topography system used as representative device for measurement of anterior corneal curvature (anterior corneal topography).

SUMMARY:
The EYESTAR 900 with software version i9.5.1.0 includes new analysis functionality. Since its clinical performance cannot be assessed based solely on clinical literature as found in the Clinical Evaluation Report, further data from a clinical trial is required. The objective of this trial is to assess the clinical performance of the new features of the EYESTAR 900 with software version i9.5.1.0.

This study is a necessary part of the clinical evaluation process of the investigational device. The results of this study are used for the clinical evaluation, and for reporting of in-vivo repeatabilities in the instructions for use of the investigational device, as required by topography standards.

DETAILED DESCRIPTION:
Ocular biometry is the act of measuring the geometric properties of the eye, in particular distances between and thicknesses of the visual axis of the cornea, lens and retina, as well as curvature of the anterior cornea. These measurements are used mainly to determine implant type and dimensions for cataract surgery.

Corneal topography is the act of measuring the shape of the cornea, in particular of the anterior cornea, but, depending on the device and the application, also of the posterior cornea, as well as the distance between the anterior to the posterior of the cornea. These measurements can be used in the context of ocular biometry, but are also useful for many other applications where knowledge of the optical and structural properties of the cornea are of interest.

Optical coherence tomography (OCT) is a well-established imaging modality in ophthalmology. It uses interferometry to obtain a scattering profile of the eye along the direction of propagation of a laser beam which is directed onto the eye. In analogy to ultrasound imaging, this scattering profile is called A-Scan. By laterally translating the measurement beam, several A-scans can be combined to form a 2-dimensional image or 3-dimensional (3D) tomogram of the eye. The main use of OCT is the cross-sectional imaging of the retina or the cornea, primarily for diagnostic purposes[4]. Recently, anterior segment OCT has also been used for corneal topography[5], as well as for biometry and cross-sectional imaging along the entire length of the eye[6].

EYESTAR 900 is a device developed by Haag-Streit which utilises 3D OCT for quantitative measurements of the geometry of the entire eye, including ocular biometry and corneal topography. CE approval for EYESTAR 900 with software version i9.4.0.0 is pending and expected before the start of this clinical trial.

The development of this device has been continued, and the following additions have been made in software version i9.5.1.0 used for this clinical study with respect to the software version i9.4.0.0:

* Extended corneal topography: corneal topography can be evaluated over an extended area (diameter of trajectory d=13mm with respect to d=8.6mm in "standard corneal topography").
* Irregularity segmentation: segmentation methods (identification of corneal surfaces) used in corneal topography now incorporate an improved algorithm for segmentation of irregular corneal surfaces.
* Irregularity visualization: visualization of topography maps has been supplemented by an overlay of regions with irregular corneal surfaces.
* Zone-based keratometry: visualization of topography maps has been further supplemented by an overlay of local keratometry values (power and axes of flat and steep meridians in the centre, middle and outer corneal surface).
* Crystalline lens tilt: the tilt of the crystalline lens normal vector with respect to the visual axis can be visualized and quantified.

Both irregularity visualization and zone-based keratometry are applicable to corneal topography data acquired with the standard corneal topography protocol, as well as corneal topography acquired over the extended area (diameter 13mm, extended corneal topography).

The primary objective of this clinical trial is to assess the clinical performance of extended corneal topography using irregularity segmentation, standard corneal topography using irregularity segmentation and crystalline lens tilt. To that end, for each measurand, the in-vivo repeatability will be quantified. For "standard corneal topography" and "extended corneal topography", the limits of agreement and the mean measurement deviation, with respect to three comparators are analyzed.

As a secondary objective of the study, raw measurement data will be collected to allow for the improvement of existing algorithms, development of additional measurands and for retrospective analysis.

Examinations with EYESTAR 900 and the other study devices are non-contact examinations. No diseases are studied as part of this study.

ELIGIBILITY:
Inclusion Criteria:

voluntary participation of subjects of legal age, irrespective of age, gender, ethnicity, of which:

* participants with healthy eyes,
* participants with corneal scarring,
* participants with irregular astigmatism.

Exclusion Criteria:

* Involuntary participation or inability to provide consent,
* persons of vulnerable populations,
* persons unable or unwilling to follow instructions,
* persons unable to maintain fixation for the duration of the examinations,
* persons with active inflammation or infections of the eye,
* persons with a tear film break up time of less than 5 sec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
In-vivo Repeatability | 3 months
  The in-vivo repeatability is calculated as the square root of the residual variance of a mixed-effects ANOVA model (using subject as a random effect, and eye within subject as a fixed effect), which we multiply with a factor of square root of two (in order to make it commensurate with the standard deviation of the differences between two independent measurements of each eye in the study sample).
  For comparator devices, the in-vivo repeatability will be assessed as well, based on two independent measurements of the same eye.
Limits of Agreement | 3 months
  For each measurand, a comparator device was defined which represents the current clinical standard. For the comparator device, for each measured parameter the mean value per eye is obtained (this value serves as the "best guess" of the true value of this parameter for one particular eye). Then, for each examination of EYESTAR 900, the difference with respect to this comparator mean value is calculated. For the resulting differences per parameter, the interval spanning the mean difference ± 1.96 * the first standard deviation of the differences is obtained. This interval quantifies the limits of agreement, spanning 95% of the expected measurement differences between EYESTAR 900 and the comparator device.
Confidence Interval of Differences | 3 months
  The mean deviation with respect to a comparator device ("equivalence") is determined as the confidence interval of a double-sided Wilcoxon test (α=0.05) of the mean measurement difference between the investigational device and the comparator device, computed over the study sample.

SECONDARY OUTCOMES:
Raw OCT Data | 3 months
  Acquisition of volumetric OCT Data of the eye. This secondary study outcome allows for the improvement of existing algorithms, development of additional measurands and for retrospective analysis but will not be processed within the scope of this clinical trial.
Raw Image Data | 3 months
  Acquisition of photographic images of the eye. This secondary study outcome allows for the improvement of existing algorithms, development of additional measurands and for retrospective analysis but will not be processed within the scope of this clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: David Goldblum, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trial ES 900 - 2019 — https://clinicaltrials.gov/ct2/show/NCT04112472